CLINICAL TRIAL: NCT04667403
Title: Telemedicine in the Management of Pain in Patients With Advanced or Metastatic Pancreatic Cancer
Acronym: PANTELO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institut Cancerologie de l'Ouest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: ICO-2020-13
Record Dates: First submitted 2020-12-01; First posted 2020-12-14 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Adenocarcinoma; Pancreatic Cancer Metastatic; Pain
Keywords: telemedicine
MeSH Terms: conditions — Adenocarcinoma; Pain | interventions — Telemedicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Telemedicine (Experimental): Pain is monitored, from the patient's home, using a computer application accessible from a smartphone or a computer with internet access.
  This application will allow the patient to describe his or her pain by means of a self-questionnaire. Healthcare professionals (nurse coordinator, pain specialist and oncologist) will thus be able to remotely interpret the data collected, enabling them to provide patients with a rapid response to adapt their pain treatment without the patient having to travel to the establishment.
  Interventions: Other: Telemedicine

INTERVENTIONS:
Other: Telemedicine — In addition to his standard follow-up, the patient benefits from a home follow-up of his pain for 6 months from his inclusion in the study.
  The patient has to log on via the application, every week. to fill in the questionnaire to evaluate the pain over the past week.
  The questionnaire consists of 4 questions to which the patient answers using a numerical scale from 0 to 10.
  If the patient's pain is not controlled, the patient can log on in "emergency" mode as many times as he or she deems necessary.
  A nurse path coordinator will be informed of each connection. Depending on the type of alert received, she may initiate a telephone consultation with the oncologist or pain specialist:
  * If necessary within 24 hours of the connection if it is a weekly connection,
  * Systematic within 3 hours if it is an emergency connection or if the data entered at the time of the weekly connection requires medical intervention.

SUMMARY:
Adenocarcinoma of the pancreas is a major public health issue because of its disastrous prognosis. The symptomatology of locally advanced or metastatic forms, particularly painful, is often major and difficult to balance, impacting both the quality of life of patients (and those around them) and the course of treatment (chemotherapy).

The objective of this study is to evaluate the interest and feasibility of telemedicine in the management of pain in patients undergoing treatment for advanced or metastatic pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 years old ;
* Patient with histologically or cytologically proven locally advanced and/or metastatic adenocarcinoma of the pancreas;
* Patient undergoing or failing medical treatment and comfort care only;
* Patient with EVA ≥ 4 and/or requiring analgesics level 3;
* Performans Status (ECOG) < 3 ;
* Informing the patient and obtaining free, informed and written consent signed by the patient and the investigator;
* Patient affiliated or beneficiary of the social security system

Exclusion Criteria:

* Patient does not have a smartphone, tablet or computer;
* Patient with no personal internet access at home (WIFI, wired), or via his smartphone;
* Patient does not feel able to fill out an electronic questionnaire;
* Patient cannot read or write French;
* Patient does not speak and understand French;
* Persons deprived of liberty or under guardianship or trusteeship ;
* Dementia, mental alteration or psychiatric pathology that could compromise the patient's informed consent and/or compliance with the protocol and follow-up of the trial ;
* Inability to submit to trial protocol follow-up for geographical, social, or other reasons ;
* Patient participating in another interventional study evaluating treatment and pain management.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-02-07 (Actual); Primary Completion 2023-11-08 (Estimated); Study Completion 2024-02-08 (Estimated)

PRIMARY OUTCOMES:
Satisfaction of patients with advanced or metastatic pancreatic cancer of the impact of telemedicine in the management of their pain. | at one month, 3 months and 6 months post-inclusion
  Satisfaction is measured using the Patient Global Clinical Impression of Change (P-GIC) questionnaire.
  The questionnaire consists of a single question posed to the patient via the application asking the patient what impact he or she believes telemedicine has had on the overall management of his or her pain. The patient has the following 8 propositions among which he must indicate the one that best corresponds to the perceived change: Don't know, Very strongly positive, Strongly positive, Slightly positive, No change, Slightly negative, Strongly negative, Very strongly negative.

SECONDARY OUTCOMES:
Observed feasibility of telemedicine | 3 months post-inclusion.
  Feasibility will be assessed by collecting :
  Number of weekly connections actually made and validated up to 3 months post -inclusion.
  Number of weekly connections actually made and not validated up to 3 months post-inclusion.
  Number of emergency connections actually made and validated up to 3 months post-inclusion.
  Number of emergency connections actually made and not validated up to 3 months post-inclusion.
  A validated connection means that the patient has answered all the questions defined for the type of weekly or emergency connection chosen and that the application has acknowledged the connection.
Satisfaction of healthcare professionals with the use of telemedicine in the management of patients' pain. | at 6 months post-inclusion
  Satisfaction is measured using the healthcare professionals Global Clinical Impression of Change (C-GIC) questionnaire. The questionnaire includes a single question asked to the medical staff taking care of the patient (Nurse pathway coordinators and oncologists or algologists) asking them to estimate the impact of telemedicine on the overall pain management of patients. They are given the following 8 propositions, among which they must indicate the one that best corresponds to the perceived change: Don't know, Very strongly positive, Strongly positive, Slightly positive, No change, Slightly negative, Strongly negative, Very strongly negative.
Number of "unscheduled" consultations recorded of each patient. | at 3 months and 6 months post-inclusion
Number of unscheduled hospitalizations recorded of each patient. | at 3 months and 6 months post-inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Julia QUINTIN, MD, Principal Investigator — Institut de Cancérologie de l'Ouest
Locations (1):
- ICO site St HERBLAIN, Saint-Herblain, France

IPD SHARING:
Plan to Share IPD: No